CLINICAL TRIAL: NCT06579846
Title: Multicenter Experimental Study to Evaluate the Efficacy in Tobacco AbstinEnce At 12 Months of DIrected Exercise and CyTisinicline
Brief Title: 12-Month Efficacy of Exercise and Cytisinicline for Tobacco Abstinence
Acronym: MEDSEC-CTA12
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Universidad de Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDSEC-CTA12
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation
Keywords: Tabacco; Cytisinicline; Exercise
MeSH Terms: conditions — Smoking Cessation; Motor Activity | interventions — cytisine; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytisinicline and exercise (Experimental): Smokers who will receive directed physical exercise and brief counseling while undergoing treatment according to the care process.
  Interventions: Drug: Cytisinicline and exercise
- Cytisinicline (Active Comparator): Smokers who will receive an informational leaflet and brief counseling when they begin cytisinicline treatment, according to the care process.
  Interventions: Drug: Cytisinicline

INTERVENTIONS:
Drug: Cytisinicline and exercise — Doctors will provide brief, personalized counseling anti-smoking plan. This counseling will support smokers in the determination-action phase of behavior change.
  Physicians will administer cytisine as follows: 1 tablet every 2 hours (maximum 6 per day) from days 1-3; every 2.5 hours (maximum 5 per day) from days 4-12; every 3 hours (maximum 4 per day) from days 13-16; every 5 hours (maximum 3 per day) from days 17-20; and 1-2 tablets per day (maximum 2 per day) from days 21-25.
  Participants will follow a combined aerobic and strength exercise program. This includes at least 150 minutes of moderate-intensity aerobic physical activity per week, or 75 minutes of vigorous-intensity aerobic activity, or an equivalent combination of both. Aerobic activity should be performed in sessions lasting at least 10 minutes.
  Other Names: Cytisinicline; Exercise
  Arms: Cytisinicline and exercise
Drug: Cytisinicline — Same intervention as the experimental group without directed exercise prescription
  Arms: Cytisinicline

SUMMARY:
Current scientific evidence demonstrates the relationship between good physical fitness and a lower incidence of certain chronic diseases, including smoking, as well as the effectiveness of cytisinicline. This protocol aims to evaluate the efficacy of the synergistic effect of combining structured physical exercise, brief counseling, and cytisinicline administration in achieving smoking cessation. The study will be an experimental, multicenter, randomized, and controlled trial with two parallel arms, conducted by a multidisciplinary team within the primary care setting of the Andalusian public health system, with a 12-month follow-up. The estimated sample size is 75 participants per arm. One of the study arms will include a structured exercise program aligned with the recently approved regional Andalusian health plan.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* Smoking a minimum of 10 cigarettes per day.
* In the contemplation or action stage according to Prochaska and DiClemente's Transtheoretical Model.
* Prepared to initiate smoking cessation treatment imminently and with commitment.
* Demonstrating a high level of nicotine dependence, with a Fagerström test score of 7 or higher.
* Exhibiting significant motivation to quit smoking, as indicated by a Richmond test score of 6 or higher.
* Having made at least one prior attempt to quit smoking within the past year.
* Enrolled in or covered by the Andalusian Public Health System.

Exclusion Criteria:

* Individuals with medical conditions that contraindicate participation in physical exercise, including but not limited to malignant hypertension, heart failure, hyperthyroidism, peripheral arterial disease, or other conditions deemed by the research team to pose a risk of adverse events or significantly impair adherence to the study.
* Individuals who have experienced changes in their usual treatment regimen within the past 90 days.
* Individuals unable to provide informed consent.
* Individuals with pathological conditions that significantly reduce life expectancy to less than 5 years.
* Individuals with contraindications as specified in the product information for cytisinicline , such as pregnancy, breastfeeding, hypersensitivity to cytisinicline, unstable angina, recent myocardial infarction, clinically significant arrhythmias, or recent stroke.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Smoking | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Number of cigarettes smoked daily.
Smoking cessation | Day 30; Day; 60; Day 90; Day 180; Day 365
  Dichotomous variable (yes/not) asking in the clinical history.
Carbon monoxide exhaled air | Day 0; Day 30; Day; 60; Day 90; Day 180; Day 365
  Carbon monoxide in the subject's exhaled air. It will be measured with a Co-oximeter of the brand "Co Check", code 01PLS18B, with a sensitivity of 1 ppm and accuracy (repeatability) of 2%. The unit of measurement of the variable is parts per million (ppm).

SECONDARY OUTCOMES:
Blood pressure | Day 0; Day 30; Day; 60; Day 90; Day 180; Day 365
  Blood pressure is measured in the non-dominant arm three times, with a 5-minute gap between each measurement, using an automatic oscillometer (Omron M3 Intellisense HEM-75051-EV; IOMRON Healthcare Europe) equipped with a child-specific cuff. The average of the three measurements is recorded for both systolic and diastolic blood pressure. The mean blood pressure values are expressed in mmHg.
Weight | Day 0; Day 30; Day; 60; Day 90; Day 180; Day 365
  Weight in grams is measured by the precision weighing scale model Tanita 780PMA.
Body mass index | Day 0; Day 30; Day; 60; Day 90; Day 180; Day 365
  Body mass index in kilograms per square meter is calculated.
Physical dependence on nicotine | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Physical dependence on nicotine measured by the Fagerström Test for Nicotine Dependence (FTND). This test consists of 6 questions, and each question has response options with assigned scores. The total score is the sum of the response scores and ranges from 0 to 10 points. The scoring scale is interpreted as follows:
  0-2 points: Low dependence. 3-4 points: Low to moderate dependence. 5 points: Moderate dependence. 6-7 points: High dependence. 8-10 points: Very high dependence.
Psychological dependence on smoking | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Physical dependence on nicotine measured by the Glover-Nilsson Smoking Behavioral Questionnaire (GN-SBQ). The GN-SBQ consists of 11 questions, each with response options ranging from 0 (never) to 4 (always), forming a 5-point Likert scale.
  The total test score is obtained by summing the responses to all the questions, resulting in a possible score range of 0 to 44 points. The scores are interpreted as follows:
  0-10 points: Low behavioral dependence on tobacco. 11-22 points: Moderate behavioral dependence. 23-33 points: High behavioral dependence. 34-44 points: Very high behavioral dependence.
Motivation to quit smoking | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Physical dependence on nicotine measured by the Richmond Smoking Withdrawal Questionnaire. This test consists of 4 questions. Each question has response options with scores ranging from 0 to 3 points. The total score is obtained by summing the responses, resulting in a possible range of 0 to 10 points.
  The interpretation of the scores is as follows:
  0-3 points: Low dependence on nicotine. 4-5 points: Moderate dependence. 6-7 points: High dependence. 8-10 points: Very high dependence.
Alcohol consumption | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Weekly alcohol consumption. Unit of measurement is Standard Drink Units
Physical activity | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Time physical activity performed daily will be measured with the Global Physical Activity Questionnaire (GPAQ) of the World Health Organization (WHO). It collects quantitative information on physical activity in three different domains:
  1) Physical activity at work (including occupational activity and domestic work); 2)Transport (physical activity related to transportation, such as walking or cycling); 3) Recreational physical activity (sports, exercise, leisure).
  For each of these domains, the GPAQ asks respondents about the frequency (days per week) and duration (minutes per day) of the physical activities performed. Additionally, the GPAQ also inquires about the time spent on sedentary activities.
  The collected information is used to calculate the respondent's level of physical activity, which is categorized into levels such as low, moderate, or high physical activity according to WHO guidelines.
Self-efficacy for physical activity | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  Self-efficacy for physical activity measured by the Benisovich Test. The scale used in this test is an 11-point Likert scale, ranging from 0 to 10, where:
  0 indicates "not confident at all" or "I have no confidence at all that I could do this." 10 indicates "completely confident" or "I have complete confidence that I could do this."
Heart rate in rest | Day 0; Day 7; Day 30; Day; 60; Day 90; Day 180; Day 365
  The unit of measure is beats per minute (bpm).

IPD SHARING:
Plan to Share IPD: No